CLINICAL TRIAL: NCT05087602
Title: Study of PD-1 Toripalimab Combined With Anlotinib in Unresectable Locally Advanced or Metastatic Acral Malignant Melanoma
Brief Title: Toripalimab Combined With Anlotinib in Unresectable Locally Advanced or Metastatic Acral Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Cuihua Yi, Director, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMM-01
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced or Metastatic Acral Malignant Melanoma
MeSH Terms: interventions — toripalimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus Anlotinib capsules (Experimental): Toripalimab 240 mg IV on Day 1 of each 14-day cycle plus Anlotinib capsules given 10mg orally in fasting conditions , once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: Toripalimab and Anlotinib

INTERVENTIONS:
Drug: Toripalimab and Anlotinib — Toripalimab 240 mg IV on Day 1 of each 14-day cycle plus Anlotinib capsules given 10mg orally in fasting conditions , once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).

SUMMARY:
Evaluate PFS of PD-1 Toripalimab Combined With Anlotinib in Subjects With unresectable locally advanced or metastatic acral malignant melanoma

DETAILED DESCRIPTION:
Malignant melanoma (MM) is one of the most malignant tumors. It is easy to metastasize at an early stage, has a high mortality rate, and its incidence is increasing year by year. This study aims to evaluate the effectiveness and safety of the combined application of Anlotinib Hydrochloride Capsules and Toripalimab in the treatment of unresectable stage III and stage IV acral malignant melanoma confirmed by pathology.

ELIGIBILITY:
Inclusion Criteria:

1.18 and 75 years; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

2.Histologically or cytologically confirmed unresectable locally advanced or metastatic acral malignant melanoma.

3.At least one measurable lesion, as defined by RECIST v1.1, that has not been irradiated. New lesions that have developed in a previously irradiated field may be used as sites of measurable disease assuming all other criteria are met.

4. Providing tumor specimen obtained by biopsy or surgical sample within 2 years 5.No prior systemic therapy or has received at least first-line treatment but appeared disease progression or intolerance.

6.The main organs function are normally. Adequate bone marrow, hepatic, and renal function documented within 4 weeks prior to treatment as documented by:absolute neutrophil count ≥ 1.5*10^9/L; platelets ≥ 100 x 10^9/ L; hemoglobin ≥ 90 g/L(no blood transfusion within 14 days before enrollment) serum creatinine ≤1.5×ULN，total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN , unless there are liver metastases in which case AST and ALT ≤5.0 x ULN;INR, aPTT, PT≤1.5 x ULN; left ventricular ejection fraction (LVEF) ≥50%. serum creatinine ≤1╳ULN，creatinine clearance >50 umol/L；urinary protein <2+ by urine dipstick. If dipstick is ≥2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours；Women of childbearing potential must have a negative serum or urine pregnancy test are received within 7 days before the randomization. Women of non childbearing age are defined as having been postmenopausal for at least 1 year, or having undergone sterilization or hysterectomy.Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 1 year after the last dose of study with an annual failure rate of less than 1% (such as intrauterine devices , contraceptives or condoms) .

7.Written and voluntary informed consent. 8.No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140, and the baseline diastolic blood pressure readings must be ≤90. Patients whose hypertension is controlled by antihypertensive therapies are eligible

Exclusion Criteria:

1. Any component of this study was not tolerated in the past.
2. Participated in other clinical trials within 4 weeks
3. Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components.
4. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks.
5. Prior therapy with VEGFR-target TKI included anlotinib or an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody ,or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways. Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of epidermoid growth factor (EGF), platelet derived growth factor (PDGF), or fibroblast growth factors (FGF) receptors.
6. Any other form of systemic or local antitumor therapy is planned for the duration of the study.
7. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration.
8. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix.
9. Has brain metastasis and cancerous meningitis during screening . Active autoimmune disease（Such as the following, but not limited to: autoimmune hepatitis interstitial pneumonia enteritis vasculitis, nephritis。Subjects with asthma requiring bronchodilators for medical intervention were not included） requiring systemic treatment（Such as the use of palliative drugs, corticosteroids, or immunosuppressants） occurred within 2 years prior to initial administration.

   Abnormal coagulation function (INR > 1.5 or PT > 1.2uln or PTT > 1.2 ULN), bleeding tendency or undergoing thrombolytic or anticoagulant therapy; treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs;
10. Has any bleeding or bleeding events ≥ grade 3 or with unhealed wounds, ulcerative , or fractures within 4 weeks prior to the first administration.
11. Received major surgical treatment or significant traumatic injury within Random 28 days prior
12. Subjects with poor blood pressure control (systolic≥ 150 mmHg or diastolic ≥100mmHg)
13. Has multiple factors affecting oral medication or malabsorption syndromes.
14. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
15. A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment. liver cirrhosis,active hepatitis*;*active hepatitis(Hepatitis B reference: HBsAg positive, and HBV DNA test value exceeds the normal valueHepatitis C reference: HCV antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value.HIV infected.
16. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first dose. Has received granulocyte colony stimulating factor(G -CSF)，or Granulocyte macrophage colony stimulating factor (GM-CSF) within 2 weeks prior to first dose
17. Subjects with a history of psychotropic substance abuse and being unable to get rid of it or with mental disord
18. Women who are pregnant or breast-feeding.
19. According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases including mental disorders need to be treated together, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | up to 2 year
  defined as the time from randomization to progress from any cause during the course of the study

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  CR+PR
Overall Survival (OS) | up to 2 year
  defined as the time from randomization to death from any cause during the course of the study
Disease control rate（DCR） | up to 1 year
  Disease control rate
Duration of overall response (DOR) | up to 1 year
  Duration of overall response

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China